CLINICAL TRIAL: NCT02784392
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Comparator-Controlled Study of the Efficacy, Safety, and Pharmacokinetics of Intravenous Ulimorelin (LP101) in Patients With Enteral Feeding Intolerance (EFI)
Brief Title: Efficacy, Safety, and Pharmacokinetics (PK) Study of Ulimorelin in Patients With Enteral Feeding Intolerance (EFI): The PROMOTE Trial
Acronym: PROMOTE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lyric Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP101-CL-201; 2016-000723-94 (EudraCT Number)
Record Dates: First submitted 2016-05-23; First posted 2016-05-27 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Enteral Feeding Intolerance (EFI)
MeSH Terms: interventions — ulimorelin; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): Ulimorelin
  Interventions: Drug: Ulimorelin
- Comparator (Active Comparator): Metoclopramide
  Interventions: Drug: Metoclopramide

INTERVENTIONS:
Drug: Ulimorelin — Active
  Arms: Active
Drug: Metoclopramide — Comparator
  Arms: Comparator

SUMMARY:
The purpose of this study is to evaluate the effect Ulimorelin in patients with enteral feeding intolerance.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, comparator-controlled study. The study consists of 2 parallel-dose treatment groups consisting of ulimorelin and metoclopramide. Approximately 120 mechanically ventilated, tube-fed patients with EFI will participate in this trial. To be eligible for study participation, the patients must be intolerant to continuous gastric tube feedings, with intolerance defined as having a gastric residual volume (GRV) of ≥ 500 mL on one or more measurements.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant women aged 18 years and above
* Intubated and mechanically ventilated in the ICU
* Receiving continuous nasogastric, orogastric, or percutaneous gastric tube feeding, with no contraindication to advancing feedings per the feeding protocol
* A 12-Fr or larger nasogastric, orogastric, or percutaneous gastric feeding tube, with its distal tip at least 10 cm below the gastroesophageal junction and visible in the stomach on a routine radiographic examination within 24 hours of screening
* Enteral feeding intolerance, defined as a GRV of ≥ 500 mL on one or more measurements Expected to remain intubated, mechanically ventilated, and receiving nasogastric feeding for at least 72 hours

Exclusion Criteria:

* Inability to obtain written informed consent to participate in the study from the patient or legally authorized representative
* Prior use during the current ICU admission of parenteral nutrition or trophic feeding, defined as a prescription to receive ≤ 20 mL/hr of enteral feeding for more than 24 hours prior to screening [N.B., parenteral nutrition may be initiated post randomization provided that the supplemental nutrition is coordinated with the calories and protein targets of the Prescribed Total Volume (PTV) and reduced as enteral feeding is advanced]
* Weight prior to ICU admission exceeding 150.0 kg
* Suspicion or confirmation of active bowel obstruction, perforation, or leakage
* History of esophageal or gastric surgery prior to or during the current hospital admission
* Use of any of the following prokinetic medications during the current ICU admission: domperidone, cisapride, neostigmine, or opioid antagonists, including alvimopan, naloxone, naltrexone, or analogs of naloxone or naltrexone; erythromycin or azithromycin [N.B., azithromycin is permitted for treatment of pulmonary infections up to 48 hours before randomization, but not thereafter through Day 5. Up to 2 doses of metoclopramide are permitted, provided that drug is not administered within 10 hours of the first dose of study drug or at any time through Day 5. If a patient receives metoclopramide during the screening period, a radiologic examination must confirm that the feeding tube remains visible in the stomach after the final dose of drug during screening and to prior to the start of baseline gastric emptying measurements and has not migrated to the duodenum. Use of clarithromycin for any indication is not excluded. Propofol must be discontinued before screening. However, its use may be permitted under special circumstances subsequent to the first dose of study drug but not in excess of 12 hours administration over the 5-day study period.]
* Patient's clinical condition is deteriorating rapidly, or the Investigator does not consider there to be a reasonable expectation that the patient will complete the study Childs C cirrhosis or Alanine Aminotransferase (ALT) ≥1000 U/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
The daily average (mean) percentage of target daily protein received through enteral nutrition by mechanically ventilated and tube-fed patients with EFI, Days 1 through 5 | 5 Days

SECONDARY OUTCOMES:
The daily average (mean) percentage of target daily calories received through enteral nutrition by mechanically ventilated and tube-fed patients with EFI, Days 1 through 5 | 5 Days

OTHER OUTCOMES:
Serious Adverse Events (SAEs) and Adverse Events (AEs), summarized by treatment group and Medical Dictionary for Regulatory Activities (MedDRA) system organ class (SOC) and preferred term. | 8 days
Clinical laboratory tests, summarized by treatment group | 6 days
Electrocardiogram (ECGs), summarized by treatment group | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: M Scott Harris, MD, Study Director — Lyric Pharmaceuticals
Locations (5):
- United States (2):
  - New Orleans, Louisiana
  - Columbus, Ohio
- Amsterdam, Netherlands
- Spain (2):
  - Barcelona
  - Madrid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.lyricpharma.com